CLINICAL TRIAL: NCT04460443
Title: Sofosbuvir Based Regimens in Treatment of COVID 19 Patients
Brief Title: Sofosbuvir in Treatment of COVID 19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sofosbuvir
Record Dates: First submitted 2020-07-04; First posted 2020-07-07 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: COVID
MeSH Terms: interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sofosbuvir and ledipsavir (Experimental): Sofosbuvir and ledipsavir plus standard of care treatment.
  Interventions: Drug: Sofosbuvir ledipsavir
- Sofosbuvir and Daklatasuvir (Experimental): Sofosbuvir and Daklatasuvir plus standard of card treatment..
  Interventions: Drug: sofosbuvir; Drug: Daclatasvir
- Standard treatment (No Intervention): Standard treatment alone

INTERVENTIONS:
Drug: sofosbuvir — Sofosbuvir once daily
  Other Names: Mpiviropack, Sovaldy, soflanork
  Arms: Sofosbuvir and Daklatasuvir
Drug: Sofosbuvir ledipsavir — Sofosbuvir ledipsavir once daily
  Other Names: mpiviropack plus
  Arms: Sofosbuvir and ledipsavir
Drug: Daclatasvir — Daklatasuvir tablets
  Other Names: daklinza
  Arms: Sofosbuvir and Daklatasuvir

SUMMARY:
Sofosbuvir containing treatment in treatment of COVID 19 Egyptian patients

DETAILED DESCRIPTION:
Sofosbuvir containing treatment of COVID 19 Egyptian patients: a randomized-controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Covid positive patients.

Exclusion Criteria:

* Contraindication to sofosbuvir or ribavirin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with response to treatment | 1 month
  The total number of patients with response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Salama, Consultant, Principal Investigator — Tanta University - Faculty of Medicine
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No